CLINICAL TRIAL: NCT02556346
Title: Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Multiple Dose Regimens of MT-3724 for the Treatment of Patients With Relapsed Chronic B-cell Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Brief Title: Pharmacokinetics (PK), Pharmacodynamics (PD), Safety, Tolerability of Multiple Dose Regimens of MT-3724 for the Treatment of Patients With Relapsed Chronic B-cell Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The patient population (CLL & SLL) was included in another ongoing study involving NHL patients.
Sponsor: Molecular Templates, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT-3724_CLL_SLL_001
Record Dates: First submitted 2015-09-16; First posted 2015-09-22 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Chronic B-cell Lymphocytic Leukemia; Small Lymphocytic Leukemia
Keywords: CD20; immunotoxin; CLL; SLL; leukemia; lymphocytic lymphoma; lymphocytic leukemia; MT-3724; relapsed; refractory; immunotherapy; cancer; antibodies; safety; pharmacokinetics
MeSH Terms: conditions — Leukemia, B-Cell; Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Lymphoid; Recurrence; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- MT-3724 Phase 1 5 mcg/kg/dose (Experimental): MT-3724 5 mcg/kg/dose IV for 6 doses over 12 days (M-W-F X 2 weeks), followed by dose escalations (Phase 1) until recommended phase 2 dose of MT-3724 is determined
  Interventions: Drug: MT-3724
- MT-3724 Phase 1 10 mcg/kg/dose (Experimental): MT-3724 10 mcg/kg/dose IV for 6 doses over 12 days (M-W-F X 2 weeks), followed by dose escalations (Phase 1) until recommended phase 2 dose of MT-3724 is determined
  Interventions: Drug: MT-3724
- MT-3724 Phase 1 20 mcg/kg/dose (Experimental): MT-3724 20 mcg/kg/dose IV for 6 doses over 12 days (M-W-F X 2 weeks), followed by dose escalations (Phase 1) until recommended phase 2 dose of MT-3724 is determined
  Interventions: Drug: MT-3724
- MT-3724 Phase 1 50 mcg/kg/dose (Experimental): MT-3724 50 mcg/kg/dose IV for 6 doses over 12 days (M-W-F X 2 weeks), followed by dose escalations (Phase 1) until recommended phase 2 dose of MT-3724 is determined
  Interventions: Drug: MT-3724
- MT-3724 Phase 1b (Experimental): MT-3724 IV for 6 doses over 12 days for up to 4 additional cycles to explore safety, tolerability and tumor response to repeat doses of MT-3724 (subject will continue with dose that was tolerated in the Phase 1 portion of the study)
  Interventions: Drug: MT-3724

INTERVENTIONS:
Drug: MT-3724 — Intravenous dosing M-W-F X 2 weeks; MT-3724 infusion over 2 hours on each dosing day over 4 week initial cycle and then 3 week repeat cycles for up to 5 total cycles.
  Arms: MT-3724 Phase 1 5 mcg/kg/dose
Drug: MT-3724 — Intravenous dosing M-W-F X 2 weeks; MT-3724 infusion over 2 hours on each dosing day over 4 week initial cycle and then 3 week repeat cycles for up to 5 total cycles.
  Arms: MT-3724 Phase 1 10 mcg/kg/dose
Drug: MT-3724 — Intravenous dosing M-W-F X 2 weeks; MT-3724 infusion over 2 hours on each dosing day over 4 week initial cycle and then 3 week repeat cycles for up to 5 total cycles.
  Arms: MT-3724 Phase 1 20 mcg/kg/dose
Drug: MT-3724 — Intravenous dosing M-W-F X 2 weeks; MT-3724 infusion over 2 hours on each dosing day over 4 week initial cycle and then 3 week repeat cycles for up to 5 total cycles.
  Arms: MT-3724 Phase 1 50 mcg/kg/dose
Drug: MT-3724 — Intravenous dosing M-W-F X 2 weeks; MT-3724 infusion over 2 hours on each dosing day over 4 week initial cycle and then 3 week repeat cycles for up to 5 total cycles.
  Arms: MT-3724 Phase 1b

SUMMARY:
This Phase I, multiple ascending dose study will seek to enroll subjects with relapsed/refractory Chronic B-cell Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL) with confirmed and measurable disease who have received standard treatment with at least one anti-CD20 antibody (e.g.; rituximab, ofatumumab) containing front-line regimen that resulted in initial response, followed by relapse/recurrence and who are not eligible for any further approved biologic therapy, chemotherapy and/or autologous stem transplantation and/or refuse alternative approved therapies and/or are unlikely to achieve clinical benefit from any therapy of higher priority by Investigator assessment.

DETAILED DESCRIPTION:
This study is intended to provide investigators and sponsor with the following information regarding the investigational new drug MT-3724 in patients with relapsed/refractory Chronic B-cell Lymphocytic Leukemia or Small Lymphocytic Lymphoma:

The maximum dose of a single course of MT-3724 given as intravenous (IV) infusions on Days 1, 3, 5, 8, 10 and 12 at which there are negligible side effects and/or at which maximum serum levels and/or at which maximum effect on blood lymphocytes are observed. Four dose levels will be investigated.

The changes in MT-3724 serum levels and blood lymphocytes over time following IV doses at different points in the study.

The changes and kinds of clinical and laboratory effects and side effects that may occur over repeated courses of MT-3724 The changes in each subject's immune status and their CLL or SLL following one or more cycles of 6 infusions.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, age 18 years or older
* Life expectancy > 3 months
* Flow cytometric confirmation of CLL is required at screening. Previous confirmation of CLL/SLL including confirmed immunohistological diagnosis with a characteristic CD5+/CD20+ B-cell immunophenotype according to WHO criteria
* For CLL: a. An absolute peripheral blood monoclonal CD20+/CD5+ B-lymphocyte count > 5000/μL for the duration of at least 3 months
* For SLL: An absolute peripheral blood monoclonal CD20+/CD5+ B-lymphocyte count < 5000/μL AND Presence of lymphadenopathy and/or splenomegaly, with histopathological evaluation of a lymph node biopsy consistent with CLL/SLL.
* Staging CLL: Rai Stage III or IV disease, or stage 0-II disease that meets NCIWG criteria for active disease requiring therapy; SLL: Intermediate or high risk by Ann Arbor Staging with Cotswald Modifications that meets criteria for active disease requiring therapy.
* Relapsed/ Refractory CLL/SLL that has progressed despite treatment with all approved therapies known to provide clinical benefit for their disease and for which the potential subject is eligible or the potential subject must have refused any other available approved treatment options prior to consideration for enrollment.
* Potential subjects must have received at least one anti-CD20 antibody containing regimen in the past that resulted in initial measurable response (partial or complete remission), followed by relapse/recurrence.
* Potential subjects for which high-dose chemotherapy and autologous stem cell transplantation (HD-ASCT) is considered a standard curative therapy are eligible for this study if the potential subject's disease has relapsed after HD-ASCT, or the potential subject is not eligible for HD-ASCT or the potential subject has refused HD-ASCT.
* Potential subjects who have had HD-ASCT must be at least 26 weeks beyond transplant.
* All potential subjects are required to have measurable disease following previous therapy for CLL/SLL. Measurable disease, as determined by NCI-WG criteria, following standard first-line or salvage therapy; this includes potential subjects with progressive disease (PDs), stable disease (SDs), or partial remission (PR) and/or Residual disease as determined by measurable disease (i.e., PDs, SDs, or PR) or by MRD positivity, determined by flow cytometry of bone marrow and/or peripheral blood (see Laboratory Manual) in potential subjects with Complete Response (CR) or CR with incomplete bone marrow recovery (CRi) (previously termed "nodular partial remission" [(nPR])
* Eastern Cooperative Oncology Group (ECOG) performance status of < 2.
* Patients must be at least 28 days past their last course of leukemia or lymphoma treatment and have recovered from side effects of such therapy completely or with only minor residual symptoms including any significant laboratory. Patients with pre-existing severe or life threatening side effects/conditions from prior therapy or due to other diseases may not be enrolled
* Female patients of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to initiating dosing. Male and female subjects with reproductive potential must agree to use acceptable contraceptive methods while on study therapy and for 12 week following their last dose of study medication.

Exclusion Criteria:

* Ongoing use of any approved or investigational anti-neoplastic therapies with the exceptions of ongoing hormonal therapy for breast cancer (without evidence of active disease) or prostate cancer (stable on hormonal therapy).
* History of an absolute anti-CD20 monoclonal antibody (MAb) refractory CLL/SLL, defined as a failure to have ever achieved a PR, CR with persistent lymphocytic nodules in the marrow ("nPR"), or CR for at least 6 months in response to at least one anti-CD20 MAb-containing regimen amongst all past CLL/SLL treatments.
* Potential subjects cannot have experienced a significant (CTCAE Grade 3 or 4 with or without neutropenia) infection within 2 weeks of the first dose of MT-3724.
* Patients who cannot comply with protocol requirements including clinic visits for intravenous infusions and birth control measures may not be enrolled.
* Female patients who are pregnant or are breast feeding.
* Patients are not eligible if they are using any other approved or investigational anti-neoplastic therapies or any other investigational therapies for any other reason.
* Patients may not be receiving systemic corticosteroid therapy at a prednisone dose > 20 mg/day (or steroid equivalent) within 2 weeks of starting study.
* Patients with uncontrolled or severe cardiovascular disease, including myocardial infarct or unstable angina within 6 months prior to start of study treatment, New York Heart Association (NYHA) Class II or greater congestive heart failure, serious arrhythmias requiring medication for treatment, clinically significant pericardial disease, or cardiac amyloidosis may not be enrolled.
* Patients with a known history of drug abuse or any chronic neurologic, psychiatric, endocrine, metabolic, immunologic, hepatic or renal disease (including a history of hemolytic uremic syndrome) that in the opinion of the Investigator would adversely affect study participation.
* Patients with known active Hepatitis C, HIV or a present history of Hepatitis B
* Patients must not have received any vaccines for 28 days prior to administration of their first dose of MT-3724 and should not receive any vaccine during the study or within 28 days after their last dose of MT-3724.
* Patients with a suspected allergy or sensitivity to any component of MT-3724 drug preparation based upon known allergies to compounds of a similar class who have had an anaphylactic or other severe infusion reaction to human immunoglobulin or monoclonal antibody administration are not eligible.
* Potential subjects who have undergone allogeneic hematopoietic stem cell transplant or any solid organ transplant.
* Autologous hematopoietic stem cell transplant within 26 weeks prior to study entry; any history of allogeneic hematopoietic stem cell transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Tolerability as measured by number of subjects with dose limiting toxicities | 28 days
  Evaluation of tolerability of MT-3724 measured by number of subjects with dose limiting toxicities (DLTs)
Safety as measured by number of subjects with Adverse Events using CTCAE | 28 days and then every 6 months for up to 24 months following first dose if subject does not continue into Phase Ib
  Safety measured by number of subjects with Adverse Events using CTCAE Version 4.03
Tolerability as measured by adverse events using CTCAE and clinical laboratory parameters | 2-3 weeks following last dose and then every 6 months for up to 24 months following first dose
  Evaluation of tolerability of MT-3724 given for up to 4 additional cycles measured by number, nature and severity of Adverse Events using CTCAE Version 4.03

SECONDARY OUTCOMES:
PK as measured by concentrations of free MT-3724 (Cmax, Cinf) | Days 1, 5, 8, 12, 23, and 28
  Evaluation of the pharmacokinetic profile of MT-3724
PK as measured by area under the curve of free MT-3724 (AUC) | Days 1, 5, 8, 12, 23, and 28
  Evaluation of the pharmacokinetic profile of MT-3724
PK as measured by time to maximum concentration of free MT-3724 ( tmax) | Days 1, 5, 8, 12, 23, and 28
  Evaluation of the pharmacokinetic profile of MT-3724
PD as measured by immunogenicity (anti-drug antibodies) | During Screening, Days 23-25, Day 1 of cycle 2, and at final end of study visit
  Evaluation of the pharmacodynamic profile of MT-3724
Tumor Response as measured by PET or CT scan | During Screening, Days 43 & 86
  Evaluation of tumor response using International Working Group Response Criteria

CONTACTS AND LOCATIONS:
Overall Officials: David Valacer, MD, Study Director — Molecular Templates